CLINICAL TRIAL: NCT00100971
Title: Dendritic/Leukemic Fusion Cell Vaccine Therapy For AML Patients In First Remission; A Phase I Clinical Trial
Brief Title: Vaccine Therapy in Treating Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol is withdrawn due to inadequate accrual
Sponsor: Boston Medical Center (Other)
Purpose: Treatment
Other Study IDs: CDR0000404382; BUMC-2003-099
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — FANG vaccine

INTERVENTIONS:
Drug: autologous tumor cell vaccine
Drug: therapeutic autologous dendritic cells
Procedure: tumor cell-derivative vaccine therapy

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells and cancer cells may make the body build an effective immune response to kill cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of autologous dendritic and leukemic fusion cell vaccine in patients with acute myeloid leukemia.
* Determine the toxicity of this vaccine in these patients.

Secondary

* Determine whether cellular immunity can be induced by this vaccine in these patients.

OUTLINE: This is a dose-escalation study.

At the time of diagnosis, patients undergo tumor cell harvest. Patients also undergo bone marrow aspiration to collect mononuclear cells to obtain dendritic cells (DC). If insufficient DCs are obtained, patients undergo leukapheresis to obtain a sufficient number of peripheral blood mononuclear cells (PBMC). The PBMC are treated in the laboratory with sargramostim (GM-CSF) and interleukin-4 for 5-7 days to produce DC. Leukemic blasts are fused to DC to generate the dendritic/leukemic fusion cell vaccine.

Patients then undergo standard induction chemotherapy to obtain a remission, followed by standard consolidation chemotherapy.

After completing consolidation chemotherapy, patients receive autologous dendritic and leukemic fusion cell vaccine subcutaneously every 2 weeks for a total of 4 doses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 patients receive escalating doses of autologous dendritic and leukemic fusion cell vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 3-9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) by bone marrow biopsy

  * Newly diagnosed
* Must have adequate dendritic cells and AML blasts isolated from bone marrow and/or peripheral blood
* No clinical evidence of CNS leukemia

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No clinically significant autoimmune disease
* No other active malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 months since prior immunotherapy

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9
Dates: Start 2004-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lerner, MD, Study Chair — Boston Medical Center
Locations (1):
- Cancer Research Center at Boston Medical Center, Boston, Massachusetts, United States